CLINICAL TRIAL: NCT06448221
Title: The Longitudinal Effectiveness of Helper of Emotional Assessment and Relationship Teaching (HEART) Smartphone- Based Videoconferencing Program in Enhancing Residents and Their Family' Health
Brief Title: Longitudinal Effectiveness of HEART Smartphone- Based Videoconferencing Program in Enhancing Residents and Family'Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202100609B0A3
Record Dates: First submitted 2024-05-24; First posted 2024-06-07 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2023-07

CONDITIONS: Communication; Health Behavior
MeSH Terms: conditions — Communication; Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RT group (Experimental): receives the RT program and uses 3 months' smartphone-based videoconferencing without the HEA system
  Interventions: Behavioral: a web-based Relationship Teaching(RT)/communication education programs
- HEART group (Experimental): receives the RT program and uses 3 months smartphone-based videoconferencing along with the HEA system
  Interventions: Behavioral: Helper of Emotional Assessment Relationship Teaching (HEART) program
- control group (No Intervention): which has only smartphone-based videoconferencing visits

INTERVENTIONS:
Behavioral: a web-based Relationship Teaching(RT)/communication education programs — receives the RT program and uses 3 months' smartphone-based videoconferencing without the HEA system.
  Arms: RT group
Behavioral: Helper of Emotional Assessment Relationship Teaching (HEART) program — receives the RT program and uses 3 months smartphone-based videoconferencing along with the HEA system
  Arms: HEART group

SUMMARY:
This study intends to understand the longitudinal effectiveness of the smartphone- based Helper of Emotional Assessment ＆Relationship Teaching (HEART) videoconferencing program in enhancing residents and family health through the employment of a sequential-methods, triangulation research design.

In the phase I lasing 18 months, it will employ: (a) a web-based RT/communication education programs which is develop based on understanding the experience of videoconferencing visit from family in nursing home, and (b) a HEA system which is for real-time face emotion recognition system used in videoconferencing will be developed and tested. In the phase II occupying the second 18 months it will evaluate the longitudinal effects of the HEART program on residents' and family's health change over time (baseline, 1 month, 3 months, and 6 months).

Nursing homes in Taiwan will be automated computerized blocked randomly assigned to three groups: (a) An RT group, which receives the RT program and uses 3 months' smartphone-based videoconferencing without the HEA system, (b) A HEART group, which receives the RT program and uses 3 months smartphone-based videoconferencing along with the HEA system, and(c) A control group, which has only smartphone-based videoconferencing visits.

ELIGIBILITY:
Inclusion Criteria:

1. residents were aged equal or higher than 60 years, resident's family were aged equal or higher than 20 years.
2. both residents and family could communicate in Mandarin or Taiwanese
3. both residents and family have no serious hearing problems
4. residents has a MMSE score equal or higher than 16 for residents with no formal education or higher than 24 for residents with at least a primary school education
5. both residents and family agree to participate,
6. family is the significant member of residents, such as caregivers.

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
family's communication knowledge | baseline, 1 month, 3 months and 6 months
  on-line test (questionnaire scored from 0 through to 100. Higher scores mean better outcome)

SECONDARY OUTCOMES:
resident health-Geriatric Depression Scale (GDS) | baseline, 1 month, 3 months and 6 months
  scale for depression( scored from 0 through to 15.Scores of 0-4 are considered normal; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.)
resident health-Activity of daily living (ADL) | baseline, 1 month, 3 months and 6 months
  assess individual's ability to perform basic self-care tasks ( (scored from 0 through to 100. higher scores mean more independence)
resident health-heart rate variation (HRV) | baseline, 1 month, 3 months and 6 months
  measurement of the variation in time between each heartbeat
resident health-profile of mood states(POMS) | baseline, 1 month, 3 months and 6 months
  scale for mood states.(scored from 0 through to 232. A lower score describing better mood state)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu Hsin Tsai, PhD, Study Chair — Chang Gung University
Locations (1):
- Catholic Mercy Hospital Attached Nursing Home, Hsinchu, Taiwan